CLINICAL TRIAL: NCT06064305
Title: Transcriptional and Proteomic Analysis of Acute Kidney Injury
Acronym: TPA-AKI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: AnIt22-03
Record Dates: First submitted 2023-09-01; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Septic AKI patients: Septic AKI patients
  Interventions: Other: No study-specific interventions
- Non-septic post-cardiothoracic AKI patients: Non-septic post-cardiothoracic surgery AKI patients
  Interventions: Other: No study-specific interventions
- non-AKI patients undergoing routine nephrectomy: non-AKI patients undergoing routine nephrectomy
  Interventions: Other: No study-specific interventions

INTERVENTIONS:
Other: No study-specific interventions — Septic AKI patients, post-cardiothoracic AKI patients and non-AKI patients undergoing routine nephrectomy. Due to the observational design of the study, no study-specific interventions are performed. The treatment of the patients is completely guided by the responsible ICU physicians and the respective specialists.

SUMMARY:
Acute kidney injury is associated with worsened outcome for critically ill patients. Sepsis-associated and non-septic cardiothoracic surgery associated AKI have been reported, nonetheless, precise pathomechanistic differences as well as detectability of transcriptional and proteomic changes in correlation with imaging and plasma markers are unclear.

DETAILED DESCRIPTION:
Acute kidney injury is a common and detrimental finding in critically ill/sepsis patients as well as non-septic patients post cardiothoracic surgery. In many cases renal replacement therapy is required and an acute kidney injury is linked to increased morbidity and mortality in intensive care patients. Using routinely obtained clinical samples as well as imaging data, this observational trial investigates the transcriptomic and proteomic determinants detectable in septic and non-septic AKI patient subsets and their correlation with outcome and AKI diagnostic parameters.

ELIGIBILITY:
* Inclusion criteria:

  * study consent;
  * KDIGO>=2;
  * vasoplegia and/or sepsis or elective nephrectomy.
* Exclusion criteria:

  * Age<18 years;
  * pregnancy/nursing;
  * preexisting CKD with eGFR<60m/min;
  * dialysis; former ogran transplantation;
  * HIV; hematologic malignancies;
  * immunsuppression;
  * 4h post biopsy non-pausable effective anticoagulation;
  * pre-existing coagulopathy

Ages: 18 Years to 150 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: AKI patients, nephrectomy patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-29 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of transcriptional and proteomic gene regulation in tissue with clinical molecular Imaging and AKI biomarkers. | Through study completion, an average of 1 year.
  Proteomic and RNAseq-based multi-omics pattern recognition.

SECONDARY OUTCOMES:
Further organ failure based on systemic assessment | Through study completion, an average of 1 year.
  Occurrence of organ failure based on hospital data including routinely applied scores, laboratory values or clinical examination.
RRT incidence | 28 days
  incidence of renal replacement therapy
ICU length of stay | Through study completion, an average of 1 year.
  Length of stay for ICU
Hospital length of stay | Through study completion, an average of 1 year.
  Hospital length of stay
Mortality | 28 day
  28 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster